CLINICAL TRIAL: NCT04153500
Title: Validation of a Female Pelvic Floor Interactive Training Model: RCT
Brief Title: Validation of a Female Pelvic Floor Interactive Training Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Autonoma de Barcelona (Other)
Responsible Party: Principal Investigator, Ana Pereda, Gynecologist, Universitat Autonoma de Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CEEAH 4764
Record Dates: First submitted 2019-10-04; First posted 2019-11-06 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Pelvic Floor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Principal investigator and the statistician will remain blind to group allocation. Outcome assessments will only be conducted by principal investigator blind to the intervention and control groups.
  Second researcher and professor will remain blind to questions included in both questionnaires: anatomy and satisfaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Methodology (No Intervention): A professor/lecturer of anatomy will carry out the session in the control group. The traditional (40 minutes total) will consist of 30 minutes of lecture (75% out of the total time), where female pelvic floor will be presented throughout theory and images. In the 2nd part, during 10 min (25%), participants will review anatomical drawings /atlases.
- Pelvic+ method (Experimental): The second researcher will carry out the session in the intervention group. The interventional session (40 minutes total) will consist of two parts: The 1st one is a lecture of 10 minutes (25% out of the total time) on female pelvic floor anatomy. In the 2nd part, during 30 min (75%), participants, in small groups of 4 people, will assemble the female pelvic floor interactive model, following the indications suggested by the second researcher. Pelvic+ is supported by an assembling manual that participants will be allowed to use.
  Interventions: Other: Anatomy class with Pelvic+ methodology

INTERVENTIONS:
Other: Anatomy class with Pelvic+ methodology — Teaching of female pelvis anatomy using a interactive training model (Pelvic+ methodology)
  Arms: Pelvic+ method

SUMMARY:
Residents increase their knowledge of female pelvis anatomy using a pelvic floor interactive model methodology (Pelvic+) compared to the traditional methodology.

DETAILED DESCRIPTION:
Objectives:

* To evaluate the residents' knowledge of the female pelvis anatomy at 3 months post intervention.
* To determine residents' satisfaction with Pelvic+ methodology compared to traditional methodology.

Material and Method:

Design: A multicentre, two arms, parallel randomized controlled trial (RCT) of an educational intervention to compare knowledge on female pelvis anatomy between Pelvic+ methodology and traditional methodology at baseline, at completion of intervention and at 3 months post-intervention.

Setting:

Teaching Unit of Midwifery of Catalonia. Institut d'Estudis Sanitaris, Barcelona, Spain.

Participants: Midwives in their 1st year of training.

Sample size: Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a two-sided test, 68 subjects are necessary in first group and 68 in the second to recognize as statistically significant a difference greater than or equal to 1.66 units. The common standard deviation is assumed to be 2.17 and the correlation coefficient between the initial and final measurement as 0.0001. It has been anticipated a drop-out rate of 20%.

Randomisation:

Prior to randomisation, consenting Teaching Unit will provide a list of their current residents' caseload. The number of participants on that caseload who meet the inclusion criteria, will be entered into the random numbers generator to create a randomly list in which to approach potential participants to intervention group or control group. Following the random list, sealed envelopes will be prepared. When the participant approach, second researcher will then seek informed consent to participate in the RCT consecutively. Once the participant has signed the informed consent to participate in the RCT, the first sealed envelope will be given to her/him sequentially.

The information contained in the sealed envelope will allocate the participant to room A or B. Being A: control group; and B: intervention group.

In situations where a participant, who had previously signed the informed consent and, before running the intervention session, decides to withdraw the study, will be removed from the RCT.

Blinding:

Principal investigator and the statistician will remain blind to group allocation. Outcome assessments will only be conducted by principal investigator blind to the intervention and control groups.

Second researcher and professor will remain blind to questions included in both questionnaires: anatomy and satisfaction.

Intervention: Pelvic+ methodology The interventional session (40 minutes total) will consist of two parts: The 1st one is a lecture of 10 minutes (25% out of the total time) on female pelvic floor anatomy. In the 2nd part, during 30 min (75%), participants, in small groups of 4 people, will assemble the female pelvic floor interactive model, following the indications suggested by the second researcher. Pelvic+ is supported by an assembling manual that participants will be allowed to use.

Control group: Traditional methodology A professor/lecturer of anatomy will carry out the session in the control group.

The traditional session will consist of 30 minutes of lecture (75% out of the total time), where female pelvic floor will be presented throughout theory and images. In the 2nd part, during 10 min (25%), participants will review anatomical drawings /atlases.

ELIGIBILITY:
Inclusion Criteria:

* midwives in their 1st year of training and who wish to participate and sign the informed consent document.

Exclusion Criteria:

1. registered midwives,
2. residents who have previously undertake another residence
3. residents who have done their Final Work Grade on pelvic floor,
4. residents who have done pelvic dissection during their grade studies
5. traditional methodology using anatomical models.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Knowledge of the female pelvis anatomy at 3 months post-intervention with Pelvic+ methodology compared to traditional methodology | 15 months
  The primary outcome of change of knowledge of the female pelvis anatomy at three months post-intervention with Pelvic+ methodology compared to traditional methodology will be measured by a self-completed questionnaire that will be completed by participants in both control and intervention groups prior to the teaching session and then three months post teaching.
  The following five anatomical topics will be researched:
  1. bone structure and obstetrical landmarks
  2. ligament structure
  3. superficial perineal muscle
  4. deep pelvis muscle
  5. nerves.
  Each of the above anatomical topics will be assessed with three questions using a Likert type scale, the total mean scores for each of the anatomical topics pre teaching and at three months post teaching for both the intervention and control groups will then be compared and analysed for comparison between the intervention and control goups.

SECONDARY OUTCOMES:
Satisfaction with Pelvic+ methodology compared to traditional methodology | 1 year
  Satisfaction with methodology: a likert-scale survey. This will consist of 12 questions with four-point agreement scale (symmetric agree-disagree scale) to measure participants agreement with a variety of statements related to the methodology of the anatomy session: theory, supporting material and time.
  All participants will be assessed to complete satisfaction questionnaire at the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Pereda, Dr, Principal Investigator — IES
Locations (1):
- Institut Estudis Salut, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No